CLINICAL TRIAL: NCT02162602
Title: Bone Mineral Accretion in Young Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of California, San Francisco (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIN-001_Bone Mineral Accretion; R01HD076321 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Bone Mineral Density Reference Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Compromised bone strength and increased fracture susceptibility pose significant morbidity and health care costs in children. Inadequate childhood bone accretion also may have lifelong consequences. Bone fragility among children with chronic medical conditions is a special concern. Identifying children at-risk for bone fragility and factors affecting bone strength requires understanding normal bone development. Dual energy x-ray absorptiometry (DXA) is the most common method for measuring bone mineral content and bone density in children. There are bone density reference data for children ages 5-20 years. An important gap is the lack of reference data for children ages < 5 years, who also experience numerous medical conditions that threaten their bone health.

Growth and body composition influence bone mineral accrual, and are important for interpreting bone density measurements in children with conditions that threaten bone health. Gross motor skills and subsequent physical activity may also affect bone accrual. Children with chronic illness are at risk of altered body composition, delayed growth and gross motor skills, and restricted physical activity. Understanding independent effects of growth, body composition, gross motor skills and physical activity on bone accrual will improve interpretation of bone density measurements and has important research and clinical applications for identifying risk factors and therapies for young children.

This study will involve a longitudinal cohort of 280 children studied every 6 months for 3 years, and a cross-sectional cohort of 240 children measured once. The study will be conducted at 2 clinical centers [Cincinnati Children's Hospital Medical Center (CCHMC) and the Children's Hospital of Philadelphia (CHOP)] with equal enrollment at both centers. Measurements will include bone density, growth and body composition, dietary intake, sleep, physical activity and gross motor skills. Results from this study will enable clinical bone health assessment of young children with disorders that threaten bone health, and identify factors that affect bone accrual.

DETAILED DESCRIPTION:
This study seeks to understand bone mineral accrual in children 1 to 5 years of age. Many young children have chronic medical conditions that threaten bone health and increase their susceptibility to fractures. Over the last 10 years our team at Cincinnati Children's Hospital Medical Center (CCHMC) has helped develop reference data that have enabled clinicians to identify children 5 to 20 y with low bone density for age and optimize their medical care. A glaring deficit is the inability to evaluate bone health of young children < 5 y due to lack of appropriate bone density reference data. This gap is problematic as there are numerous clinical conditions (e.g., neuromuscular disease, cancer, glucocorticoid treatment, extreme prematurity) that threaten bone health in this young age group.

The primary goal of our new study is to develop bone mass and density reference data to aid identification of children 1 to 5 years of age with bone deficits. A first step is to characterize the age-related changes in bone accrual at multiple skeletal sites and determine when sex and race differences in bone mass and density emerge.

The second goal of this study is to assess the influence of growth, body composition, gross motor skills and physical activity on bone mineral accrual in young children. In older children, the need to account for growth and lean mass when interpreting bone measurements has been demonstrated. The best way to do this in young children is unknown. Pronounced changes in gross motor skills, locomotion and physical activity also occur during early childhood. It is well appreciated that mechanical loads on the growing skeleton promote bone mineral accrual. but how gross motor skills and physical activity impact bone development in children 1 to 5 years of age is unknown. Understanding the impact of growth, body composition, motor skill development, and physical activity on bone accrual in young children is important for interpretation of clinical bone density measurements. These characteristics are often affected in young children with chronic medical conditions.

This study will enroll 520 healthy children between 1 to 5 years of age; half will be recruited at CCHMC and half at Children's Hospital of Philadelphia.

This study is unique since no previous studies have addressed these issues in children 1-5 y. It is clinically relevant as findings will facilitate medical care of children with chronic medical conditions that threaten bone health, and it will develop and validate novel methods for bone and body composition assessment in this age range. It will also add generalizable knowledge to enhance understanding of the growing skeleton, and its relationship to motor and somatic development. Since poor bone mineral accrual can have lifelong consequences, this study addresses the major public health concern of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll healthy, normally growing children free from medical conditions that may affect bone or growth between the ages of 1-5 years.

Exclusion Criteria:

* Weight, length and weight-for-length outside ± 2 Standard Deviations of the 2006 World Health Organization growth standard for ages 1 to 2 y and the 3rd to 97th percentiles of the Centers for Disease Control 2000 growth reference for ages ≥ 2 years as recommended;84 chronic medical conditions affecting bone density (e.g., cancer, kidney, gastrointestinal, musculoskeletal or endocrine disorder); chronic use of medications that affect bone (glucocorticoids, anti-epileptics, or hormones); prior fracture; dietary restrictions; preterm birth (<37 wk gestation) and low birth weight (<2500 g).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2014-05; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Baseline

SECONDARY OUTCOMES:
Bone mineral content | Baseline

OTHER OUTCOMES:
Change in bone mineral density | Over 3 years
Change in bone mineral content | Over 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Kalkwarf, PhD, Principal Investigator — Cincinnati Children's; Babette Zemel, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania